CLINICAL TRIAL: NCT00032838
Title: The Effects of Cortisol and Norepinephrine Modulation on Emotional and Nonemotional Processing
Brief Title: Effects of Stress Hormones on Emotion and Cognition
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020155; 02-M-0155
Record Dates: First submitted 2002-04-03; First posted 2002-04-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Healthy
Keywords: Hydrocortisone; Yohimbine; Cognition; Norepinephrine; Cortisol; Emotion; Healthy Volunteer; HV; Normal Control
MeSH Terms: interventions — Yohimbine

INTERVENTIONS:
Drug: Yohimbine

SUMMARY:
The purpose of this study is to examine how hormonal changes that occur during stressful situations affect thought and emotions. Results from this study may lead to treatments that can alleviate the psychological effects of trauma.

Levels of cortisol and norepinephrine increase in response to stress; these hormones also influence thought processes. This study will give hydrocortisone and/or yohimbine (a stimulator of central norepinephrine) to healthy adults in order to model the stress response and to better understand the way people process information during traumatic events.

This study comprises two experiments in which the stress response is pharmacologically modeled. Participants in the study will have two study visits. During Visit 1, participants will undergo a psychiatric assessment, complete neuropsychological tasks, and have their IQ measured. During Visit 2, participants will be given hydrocortisone and/or yohimbine. Blood will be collected before and during this. Participants will then perform two experiments. In one experiment, participants will hear a story with emotional and non-emotional segments; in a second experiment, participants will view both emotional and non-emotional stimuli.

DETAILED DESCRIPTION:
Memories for traumatic events are fundamentally different from typical memories. Individuals who witness or are involved in an extremely stressful event, such as a robbery or a violent act, retain highly accurate memories for the information directly related to the trauma (e.g., a gun or verbal threat), while surrounding details are poorly remembered. This so-called weapon focus phenomenon has been found in both naturalistic and laboratory studies with humans. However, difficulties with the control of naturalistic studies and approximating trauma in the lab limit the validity of these findings.

Neurophysiologically, cortisol and norepinephrine are principal mediators of the stress response, and both influence memory function. In particular, cortisol improves memory at low levels but impairs memory at higher doses. Similarly, some evidence indicates that norepinephrine also enhances memory in low doses and either impairs or does not influence memory at high doses. Much of the experimental work in this area has been conducted with animals. Studies have recently begun to extend these paradigms to humans.

To better understand memory processing during trauma, hydrocortisone and/or yohimbine (a stimulator of central norepinephrine) will be administered to healthy adults in two experiments in order to pharmacologically model the stress response. Following infusion, participants will hear a story with emotional and nonemotional segments in one experiment (N = 80) and emotional as well as nonemotional stimuli (faces and scenes) in another experiment (N = 80). It is predicted that relative to the placebo, hydrocortisone will impair memory for both emotional and nonemotional information, yohimbine will improve memory for both types of information, and the combination of hydrocortisone and yohimbine will enhance memory for emotional aspects and impair memory for the nonemotional segments of the story. Results from this study will permit a better understanding of how emotionally charged memories are encoded and will potentially lead to treatments to mitigate the psychological effects of traumatic exposure.

ELIGIBILITY:
INCLUSION CRITERIA:

Age: 18-36

IQ: all subjects will have IQ greater than 85

Follicular cycle: Women will participate in the encoding task between days 3-10.

EXCLUSION CRITERIA:

Pregnancy/Nursing

Only healthy individuals will participate; special attention will be taken to ensure that no subject has: hypertension, glaucoma, cataracts, ulcers, renal insufficiency, osteoporosis, hypothyroidism, cirrhosis, ocular herpes simplex and myocardial infarction.

Use of hormonal contraception

Use of glucocorticoids within past 3 years

Use of any psychoactive substance; current or past psychiatric diagnosis.

Irregular sleep pattern as defined as getting less than 6 hours of sleep per night, going to sleep after 2:00 AM; waking up before 5:00 AM or after 11:00 AM

Weight that is 15% more or less than ideal body weight for sex and height

History of panic attacks or first degree relative with history of panic attacks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170
Dates: Start 2002-03; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Diamond DM, Fleshner M, Ingersoll N, Rose GM. Psychological stress impairs spatial working memory: relevance to electrophysiological studies of hippocampal function. Behav Neurosci. 1996 Aug;110(4):661-72. doi: 10.1037//0735-7044.110.4.661. PMID 8864259
- [Background] Sandi C, Loscertales M, Guaza C. Experience-dependent facilitating effect of corticosterone on spatial memory formation in the water maze. Eur J Neurosci. 1997 Apr;9(4):637-42. doi: 10.1111/j.1460-9568.1997.tb01412.x. PMID 9153570
- [Background] Christianson SA, Fallman L. The role of age on reactivity and memory for emotional pictures. Scand J Psychol. 1990;31(4):291-301. doi: 10.1111/j.1467-9450.1990.tb00841.x. PMID 2274761